CLINICAL TRIAL: NCT03907202
Title: A Double-blind, Placebo-controlled, Randomised, Multiple-ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of KBP-089 in Patients With Type II Diabetes
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability, PK, PD, and Efficacy of KBP-089 in Patients With T2DM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was planned to be conducted in 4 cohorts but was terminated after completion of Cohort 2 for strategic reasons due to limited PD effects.
Sponsor: KeyBioscience AG (Industry)
Collaborators: Eli Lilly and Company (Industry); Nordic Bioscience A/S (Industry); Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KBP089/CD/002
Record Dates: First submitted 2018-04-17; First posted 2019-04-08 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Type II Diabetes Mellitus
Keywords: Sub-cutaneous injection; Metformin; KBP-089; randomised; placebo-controlled; multiple-ascending dose
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomised, patient-blind, investigator-blind, placebo-controlled, multiple ascending dose study. There will be 3 cohorts in which patients are randomised to receive either treatment with KBP-089 or placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: To preserve the blinding of the study for KBP-089 and placebo, all study site personnel, except pharmacy staff who prepare and dispense study medication, and the Sponsor's medical monitor who interacts with site personnel will be blinded to treatment allocation. Blinding of KBP-089 and placebo will be maintained throughout the conduct of the trial until after the completion of the trial and final data review.
  Treatment assignment will be kept strictly confidential and accessible only to authorised persons until after the time of unblinding. Codes with treatment assignment will, however, be readily available to the blinded personnel in case of an emergency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KBP-089 (Active Comparator): Three cohorts:
  * Cohort 1: starting dose 5 µg, maximum dose 20 µg, uptitration step 7 days, dose increment 5 µg
  * Cohort 2: starting dose 7.5 µg, maximum dose 60 µg, uptitration step 3 days, dose increment 7.5 µg
  * Cohort 3: starting dose 5 µg, maximum dose 120 µg, uptitration step 3 days, dose increment 5, 10, 15 and 20 µg
  Interventions: Drug: Daily injection of KBP/placebo for up to 28 days
- Placebo (Placebo Comparator): For all the cohorts, sentinel dosing for the first two patients will be performed 1:1 in a blinded manner.
  Interventions: Drug: Daily injection of KBP/placebo for up to 28 days

INTERVENTIONS:
Drug: Daily injection of KBP/placebo for up to 28 days — Daily sub-cutaneous injection of KBP-089/Placebo into a lifted skin fold of the abdominal wall.The injection will be administered in the morning before breakfast.

SUMMARY:
KeyBioscience is developing KBP-089, a dual activator of both the amylin and calcitonin receptors, for the treatment of type II diabetes mellitus, using a subcutaneous injectable mode of administration.

This is a double-blind, placebo-controlled, randomised, multiple-ascending dose phase I trial to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of KBP-089 in patients with type 2 diabetes, who are on stable therapy with metformin.

Subjects will receive daily subcutaneous injections in the abdomen over a period of 28 days. The planned maximum doses of KBP-089 to be investigated in the trial are 20 µg in cohort 1, 60 µg in cohort 2, and 150 µg in cohort 3. For cohort 1, the dose is planned to be escalated every 7 ±1 days, and for cohort 2 and cohort 3, every 3 days. Doses may be modified according to individual tolerability, but the dose regimen will not exceed 28 days.

The IMP is administered by daily subcutaneous injections taken in the morning before breakfast.

The trial is performed in Germany and at least 36 patients will be enrolled in the trial. The trial will be randomised 1:1:1 between maximum doses of KBP-089 of 20 µg, 60 µg, 150 µg and placebo. Within each of the three cohorts, 12 patients will be randomised 3:1 to KBP-089 and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedures that would not have been performed during normal management of the patient).
* Male or female patient with T2DM.
* Age between 18 and 64 years, both inclusive.
* Body Mass Index (BMI) >= 25.0 kg/m^2.
* HbA1c >= 7 and <=9.5%.
* Stable therapy with metformin ± treatment with a second oral anti-diabetes drug (OAD) belonging to the class of dipeptidyl-peptidase 4 (DPP-4) inhibitors or sulfonylureas for at least 2 months prior to inclusion into the trial or not treated with glucose-lowering medications. Patients who are receiving stable treatment with a second OAD will be asked to discontinue the DPP-4 inhibitor or a sulfonylurea for at least 14 days prior the Initial Inpatient Dosing Visit.
* Considered generally healthy (apart from T2DM) upon completion of medical history, physical examination, vital signs, ECG and analysis of laboratory safety variables, as judged by the Investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity or allergy to paracetamol or related products.
* Prior treatment with a dual amylin and calcitonin receptor agonist (DACRA) or salmon calcitonin.
* Receipt of any medicinal product in clinical development within 30 days or 5 half-lives of the medicinal product (whichever is longer) before randomisation in this trial.
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
* Any history or presence of clinically relevant cardiovascular, pulmonary, respiratory, gastrointestinal, hepatic, renal, metabolic, endocrinological (with the exception of conditions associated with diabetes mellitus), haematological, dermatological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynaecologic (if female), or infectious disease, or signs of acute illness as judged by the Investigator.
* Medically unable or unwilling to discontinue current anti-diabetic therapy with DPP-4 inhibitor or sulfonylurea for at least 14 days prior to admission to the research facility (Day -2) and remain off medication until the follow-up visit. Patients taking metformin therapy at entry will continue their metformin at the usual individual dose throughout the trial.
* Have had a significant change in weight, defined as a gain or loss of at least 5% body weight in the 3 months prior to screening.
* A positive result in the alcohol and/or urine drug screen at the screening visit.
* Positive to the screening test for Hepatitis Bs antigen (HBsAg) or Hepatitis C antibodies and/or a positive result to the test for human immunodeficiency virus (HIV)-1/2 antibodies or HIV-1 antigen.
* Have had a blood transfusion or severe blood loss within the past 6 months or have known hemoglobinopathy, hemolytic anemia, sickle cell anemia, or have a hemoglobin value <11 g/dL (males) or <10 g/dL (females), or any other condition known to interfere with HbA1c methodology.
* Blood donation or blood loss of more than 500 mL within the last 3 months or any blood donation within the last month prior to screening.
* Females of childbearing potential.
* Males with pregnant partners.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs). | Day -1 to day 28
  All TEAEs will be coded using MedDRA and summarized by treatment and dose.
Vital sign - Blood Pressure. | Day -1 to day 28
  Diastolic and systolic blood pressure (mmHg) are measured after at least 5 min rest in a supine position.
  Vital signs will be summarised by descriptive statistics by treatment, dose and timepoint.
Vital sign - Pulse (beats per min). | Day -1 to day 28
  measured after at least 5 min rest in a supine position. Vital signs will be summarised by descriptive statistics by treatment, dose and timepoint.
Vital sign - Body Temperature. | Day -1 to day 28
  Body temperature, tympanic (in Celcius). Vital signs will be summarised by descriptive statistics by treatment, dose and timepoint.
Vital sign - Respiratory frequency. | Day -1 to day 28
  Respiratory frequency measured as breaths per min. Vital signs will be summarised by descriptive statistics by treatment, dose and timepoint.
Electrocardiogram (ECG) - PQ interval. | Day -1 to day 28
  PQ interval (in msec) and any abnormality will be recorded and described in the CRF including the Investigator's assessment of clinical significance ('abnormal, not clinically significant' or 'abnormal, clinically significant').
Electrocardiogram (ECG) - QRS complex. | Day -1 to day 28
  QRS interval (in msec) and any abnormality will be recorded and described in the CRF including the Investigator's assessment of clinical significance ('abnormal, not clinically significant' or 'abnormal, clinically significant').
Electrocardiogram (ECG) - QT interval. | Day -1 to day 28
  QT interval (in msec) and any abnormality will be recorded and described in the CRF including the Investigator's assessment of clinical significance ('abnormal, not clinically significant' or 'abnormal, clinically significant').
Safety laboratory parameter - lipids. | Day -1 to day 28
  Standard Lipid assessments will be summarized by treatment (including dose) using descriptive statistics (number, mean, standard deviation, minimum, median and maximum).
  (Lipid parameters measured: Total cholesterol, High-density lipoprotein (HDL) cholesterol, Low-density lipoprotein (LDL) cholesterol, Triglycerides).
Safety laboratory parameter - haematology. | Day -1 to day 28
  Standard Biochemistry assessments will be summarized by treatment (including dose) using descriptive statistics (number, mean, standard deviation, minimum, median and maximum).
  (Haematology parameters measured: Haematocrit, Haemoglobin, Erythrocytes, Mean corpuscular volume (MCV), Mean corpuscular haemoglobin (MCH), Mean corpuscular haemoglobin concentration (MCHC), Thrombocytes (platelets), Leucocytes, Neutrophile granulocytes (total count and relative), Lymphocytes (total count and relative), Monocytes (total count and relative), Eosinophile granulocytes (total count and relative), Basophile granulocytes (total count and relative))
Safety laboratory parameter - coagulation. | Day -1 to day 28
  Standard coagulation assessments will be summarized by treatment (including dose) using descriptive statistics (number, mean, standard deviation, minimum, median and maximum).
  (coagulation parameters measured: International normalised ratio (INR), Activated partial thromboplastin time (APTT)
Safety laboratory parameter - urinalysis. | Day -1 to day 28
  Standard Biochemistry assessments will be summarized by treatment (including dose) using descriptive statistics (number, mean, standard deviation, minimum, median and maximum).
  (Urinalysis parameters measured: Protein, Glucose, Erythrocytes, Leucocytes, pH, Ketones)

SECONDARY OUTCOMES:
Pharmacokinetic Evaluation - KBP-089 Area Under Curve. | Day -1 to day 28
  PK parameter (AUC 0-24) will be derived by non-compartmental analysis of the plasma concentration data for KBP-089
Pharmacokinetic Evaluation - KBP-089 Cmax. | Day -1 to day 28
  PK parameter (Cmax) will be derived by non-compartmental analysis of the plasma concentration data for KBP-089
Gastric emptying - Paracetamol Cmax. | Day -1 to day 28
  Gastric emptying is measured using paracetamol Cmax at baseline (Day -1), Day 1, and Day 28 for Cohorts 1 and 2 only
Gastric emptying - Paracetamol Tmax. | Day -1 to day 28
  Gastric emptying is measured using paracetamol Tmax at baseline (Day -1), Day 1, and Day 28 for Cohorts 1 and 2 only
Gastric emptying - Paracetamol Area Under Curve (AUC). | Day -1 to day 28
  Gastric emptying is measured using paracetamol AUC at baseline (Day -1), Day 1, and Day 28 for Cohorts 1 and 2 only
Fasting and postprandial glucose concentration. | Day -1 to day 28
  Fasting and postprandial glucose following OGTT at baseline (Days -1) and Day 28
Fasting and postprandial insulin concentration. | Day -1 to day 28
  Insulin following OGTT at baseline (Days -1) and Day 28
Fasting and postprandial C-peptide concentration. | Day -1 to day 28
  Fasting and postprandial C-peptide following OGTT at baseline (Days -1) and Day 28
Fasting and postprandial glucagon concentration. | Day -1 to day 28
  Fasting and postprandial glucagon following OGTT at baseline (Days -1) and Day 28
Body weight. | Day -1 to day 28
  Body weight at Day -1 (baseline) and Day 28 (in kg)
N-(1-deoxy)-fructosyl-haemoglobin (HbA1c). | Day -1 to day 28
  HbA1c at Day -1 (baseline) and Day 28 (in mmol/mol)
Fridericia's corrected QT interval (QTcF). | Day 1 to day 27
  Fridericia's corrected QT interval (QTcF) at Day 1 and Day 27 (in msec)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Undecided